CLINICAL TRIAL: NCT06270186
Title: Feasibility of a Virtual Reality Approach in the Assessment of Executive Functions in Patients With Type 1 Myotonic Dystrophy : Pilot Study
Brief Title: Evaluation of Cognitive Functions in 20 Patients With Type 1 Myotonic Dystrophy With Virtual Reality Approach
Acronym: GoodDiagNMD
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: study withdrawn by the sponsor for logistical reasons
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 20-AOIP-04
Record Dates: First submitted 2022-01-14; First posted 2024-02-21 (Actual); Last update posted 2024-02-21 (Actual); Status verified 2024-02

CONDITIONS: Myotonic Dystrophy 1
MeSH Terms: conditions — Myotonic Dystrophy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Type 1 myotonic dystrophy (Other): Type 1 myotonic dystrophy patients doing classical neuropsychological test and on "Good Diag NMD" software
  Interventions: Diagnostic Test: Type 1 myotonic dystrophy

INTERVENTIONS:
Diagnostic Test: Type 1 myotonic dystrophy — To compare classical neuropsychological test and on "Good Diag NMD" software in Type 1 myotonic dystrophy patients

SUMMARY:
Type 1 myotonic dystrophy (MD1) is a genetic and hereditary disease that primarily affects muscle tissue, resulting in myotonia (difficulty relaxing after contraction) and atrophy (progressive muscle weakening with decreased muscle volume). It also affects eyes, heart, endocrine system, gastrointestinal system and central nervous system. Specific cognitive abilities are impaired in patients with MD1 such as attention, visio-spatial or visio-building abilities as well as executive dysfunctions.

Currently, the cognitive assessment of MD1 patients is based on classical neuropsychological tests, which are time-consuming and require a MD1 expert neuropsychologist. Moreover, it is usually very difficult for MD1 patients to accept performing these tests, and when they agree to perform them, they usually give up before the end. This finding is more frequent in MD1 patients with high level of cognitive impairment.

In order to overcome these difficulties in assessing cognitive functions of MD1 patients, the investigators decided to use innovative tools such as virtual reality, which allow individuals to experience a sensory-motor and cognitive experience in a digitally world through a helmet, glasses and joysticks.

The start-up My Cyber Royaume from Lille, in collaboration with the reference center of neuromuscular diseases from Nice coordinated by Pr Sacconi, have developed a software "Good Diag NMD" which uses virtual reality to assess cognitive disorders, more specifically executive functions in patients with type 1 myotonic dystrophy.

ELIGIBILITY:
Inclusion Criteria:

* male or female age ≥ 18
* suffering with type 1 myotonic dystrophy confirmed by molecular biology
* suffering with dysexecutive impairments, with a pathologic BREF score ≤ 15
* affiliated to social security
* able to understand the inform consent form

Exclusion Criteria:

* suffering with visual or auditive impairments preventing them doing tests
* suffering with other pathologies preventing them doing tests
* suffering with motor impairments preventing them holding joysticks or carrying helmet
* protection by law under guardianship, or who cannot participate in a clinical study under Article L. 1121-16 of the French Code of Public Health
* patient under treatment that may affect cognitive functions (ie : Modafinil)
* participation in the last 3 months in a clinical research study in which he / she has been exposed to a pharmaceutical product or a medical device
* pregnant or breastfeeding female patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-11 (Estimated); Primary Completion 2024-11 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
Evaluate the feasibility of the use "Good Diag NMD" software in the evaluation of cognitive executive dysfunctions in patients with dystrophy myotonia 1 | 0 months
  The feasibility "Good Diag NMD" software in patient with type 1 myotonic dystrophy (DM1) will be determined as the rate of patients having completed the Good Diag NMD session in full. Satisfactory feasibility is considered if this rate of patients is greater or equal to 50%.

SECONDARY OUTCOMES:
Establish a possible relationship between the genotype of DM1 patients and the scores obtained during "Good Diag NMD" session | 0 months
  Genotype of DM1 patients will be determined by molecular biology technique, ie the size of GTC triplet expansion will indicate the of severity of the genetic abnormality . Then, we will analyse a possible correlation of the genotype with the scores obtained during "Good Diag NMD" session.
To compare the satisfaction score of type 1 myotonic dystrophy patients between classic neuropsychological tests and the Good Diag NMD session | 0 months
  The satisfaction will be measured with a satisfaction questionnaire called "Assessment questionnaire" (value between 0 to 50)
Compare the scores of "Good Diag NMD" session (scores of perseveration, inhibition and flexibility) with the scores of the classical neuropsychological tests | 0 months
  The following correlations will be examined studied:
  * The level of correlation between perseveration score (0-149) and Frontal Efficiency Rapid Battery (BREF) score (0-18)
  * The perseveration score (0-149) and Short Cognitive Battery (B2C) score
  * The inhibition score (0-77) and interference score (score I) from Stroop test (-30 and +30)
  * flexibility score (0-119) and completion time of Trail Making Test (TMT) B
Establish a possible correlation between the severity of the disease, the severity of muscular impairment and the scores of Good Diag NMD session | 0 months

CONTACTS AND LOCATIONS:
Overall Officials: Sabrina SACCONI, Principal Investigator — Centre Hospitalier Universitaire de Nice

IPD SHARING:
Plan to Share IPD: No